CLINICAL TRIAL: NCT04731233
Title: A Randomized, Double-Blind Study of the Efficacy of Platelet-Rich Growth Factor (PRGF) Supplementation Compared to Steroid Supplementation After Temporomandibular Joint (TMJ) Arthrocentesis in Female Patients With TMJ Osteoarthritis (OA)
Brief Title: Efficacy of PRGF Supplementation After TMJ Arthrocentesis in Patients With TMJ Osteoarthritis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Could not recruit participants due to their refusal to be randomized in the study.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202000689-A; OCR40106 (Other: UF OnCore)
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: TMJ; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Intercellular Signaling Peptides and Proteins; Dietary Supplements; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PRGF Arm (Experimental): The PRGF experimental group will have two cc of PRGF infused into the upper joint space after the TMJ arthrocentesis procedure.
  Interventions: Biological: Plasma Rich in Growth Factor (PRGF) Supplementation
- Steroid Arm (Active Comparator): Two cc containing 40 mg of triamcinolone acetonide with 5 mg bupivacaine will be infused into the upper joint space after the TMJ arthrocentesis procedure.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Biological: Plasma Rich in Growth Factor (PRGF) Supplementation — After rinsing the joint, the TMJ will be injected with blood plasma rich in growth factors (PRGF). PRGF supplementation which is an autologous platelet-enriched plasma obtained from patient's own blood, which after activation with calcium chloride allows the release of a pool of biologically active proteins that influence and promote a range of biological processes.
  Arms: PRGF Arm
Drug: Triamcinolone Acetonide — After rinsing the joint, the TMJ will be injected with 40 mg of triamcinolone acetonide with 5 mg bupivacaine.
  Other Names: Kenalog
  Arms: Steroid Arm

SUMMARY:
Temporomandibular joint (TMJ) osteoarthritis (OA) affects articulating tissues secondary to inflammation resulting in intracapsular pain. This prospective, double-blind randomized clinical trial will evaluate the relative efficacy of TMJ arthrocentesis with a supplementation of platelet-rich growth factors (PRGF) compared to TMJ arthrocentesis with a steroid supplementation (a known effective therapy) for patients with TMJ OA.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMD) are musculoskeletal disorders that are commonly encountered, with pain in the temporomandibular joint (TMJ) and jaw closing muscles. Pain that involves the temporomandibular joint includes inflammatory pathologies such as arthritides, painful disk displacements and many times have an overlay of psychosocial comorbidities due to the uncontrolled pain. TMJ osteoarthritis is an intracapsular condition affecting the temporomandibular joint and presents with remodeling of the TMJ articulating tissues including the condyle and articular eminence secondary to inflammation resulting in intracapsular pain. There is a paucity of information regarding the relative effectiveness of different therapies for the treatment of patients with TMJ osteoarthritis. The identification of the least invasive and most efficacious therapy is vital to proper management of these patients with temporomandibular joint pain and disability. The purpose of this study is to establish the relative efficacy of TMJ arthrocentesis with steroid supplementation (a known effective therapy) compared to TMJ arthrocentesis with a supplement of plasma rich in growth factors (PRGF) for patients with TMJ osteoarthritis. Plasma rich in growth factors is isolated from the patient's own blood and injected into the temporomandibular joint to activate stem cells that may restore some of the articulating tissues that were lost during degeneration changes within the joint secondary to osteoarthritis. Pain and disability will be assessed using standard pain and physical measures that are recorded before and after treatment. Patients enrolled into the study will be examined and treated at the Department of Oral and Maxillofacial Surgery Faculty/Resident clinic. At the first appointment, they will be examined following standard procedures (medical history, physical exam, imaging by cone beam computerized tomography (CBCT)) to determine their diagnosis(es) and if they would potentially benefit from the TMJ arthrocentesis procedure. If the patient meets the inclusion criteria for the study and with their informed consent on the day of their TMJ arthrocentesis procedure, they will be required to have a pregnancy test if below age 60 and complete a questionnaire about their physical and pain symptoms and undergo a standardized clinical exam. The patients will then undergo the standard clinical protocol for TMJ arthrocentesis followed by either a 2 cc steroid/bupivacaine hydrochloride supplementation (standard treatment group) or a 2 cc PRGF supplementation (experimental group) into the TMJ. Follow-up appointments will be conducted at 1 month, 3 months and 6 months when the pain VAS measures and a clinical exam will be assessed. If patients have not experienced improvement in their primary outcome measure (TMJ pain) at the 3 month evaluation, the patient will have a second TMJ arthrocentesis procedure that will be supplemented with the alternative medication/growth factors (steroid or PRGF) using a cross-over design. Data from these patients will be analyzed separately from patients that complete the six month study. Also at 6 months, a second CBCT image of the temporomandibular joints will be obtained to determine the extent of bone remodeling within the TMJ. The results of this study should provide new information on the efficacy of PRGF supplementation for management of temporomandibular joint osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 40 - 80 years of age
* Unilateral or bilateral TMJ arthralgia
* Osteoarthritis diagnosis according to the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD)
* TMJ sounds (crepitus or click or both)
* Mild-moderate masticatory muscle myalgia
* History of non-surgical treatment for at least 6 weeks including such modalities as appliance therapy, NSAID therapy or physical modalities without resolution of pain

Exclusion Criteria:

* Contraindication to sedation including pregnancy or medical history
* Rheumatologic disorders causing arthritis of the temporomandibular joint (i.e., rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis)
* History of previous TMJ procedure including arthrocentesis, arthroscopy or arthrotomy
* History of steroid injection in TMJ
* TMJ pain greater than five years
* History of narcotic drug use on a scheduled basis
* Current active infection
* Fibromyalgia

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females will be studied since greater than 95% of the patients that pursue temporomandibular joint arthrocentesis are female.
Enrollment: 5 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles G. Widmer, DDS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 02-17-2021 to 02-21-2024 Study location: Oral and Maxillofacial Surgery Clinic
Period: Overall Study
Arm/Group | PRGF Arm | Steroid Arm
Started | 4 | 1
Completed | 4 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRGF Arm | Steroid Arm | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 | 5
Temporomandibular Joint (TMJ) Intracapsular Pain-Visual Analog Scale (VAS) Rating [Mean (Standard Deviation); unit: units on a scale] — The Visual Analog Scale (VAS) is a pain rating scale that has a range of 0-100 and is represented as a 100 mm line. On this scale, 0 is represented as "no pain" and 100 is represented as "the most intense pain imaginable". Pain is measured by having the subject place a line bisecting a 100 mm line to represent the pain level and a numerical rating is obtained by measuring the distance, in mm, from the zero-pain anchor (left side of scale represented by 0 pain).
  units on a scale | 67.5 (27.5) | 90.0 (0.0) | 78.6 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Temporomandibular Joint (TMJ) Visual Analog Scale (VAS) Pain Rating
Description: The Visual Analog Scale (VAS) is a pain rating scale that has a range of 0-100 and is represented as a 100 mm line. On this scale, 0 is represented as "no pain" and 100 is represented as "the most intense pain imaginable". Pain is measured by having the subject place a line bisecting a 100 mm line to represent the pain level and a numerical rating is obtained by measuring the distance, in mm, from the zero-pain anchor (left side of scale represented by 0 pain).
Time Frame: Three Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRGF Arm | Steroid Arm
Number analyzed (Participants) | 4 | 1
units on a scale | 25.0 (50.0) | 90.0 (0.0)

2. Primary Outcome: Temporomandibular Joint (TMJ) Visual Analog Scale (VAS) Pain Rating
Description: as for outcome 1
Time Frame: Six Months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | PRGF Arm | Steroid Arm
Number analyzed (Participants) | 4 | 1
units on a scale | 0.0 (0.0) | 80.0 (0.0)

3. Other Pre Specified Outcome: Chewing Pain Measured by Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRGF Arm | Steroid Arm
Number analyzed (Participants) | 4 | 1
units on a scale | 80.25 (11.7) | 78.6 (10.8)

4. Other Pre Specified Outcome: Chewing Pain Measured by Visual Analog Scale (VAS)
Description: as for outcome 1
Time Frame: Six Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRGF Arm | Steroid Arm
Number analyzed (Participants) | 4 | 1
units on a scale | 2.25 (4.5) | 42 (0.0)

5. Other Pre Specified Outcome: Temporomandibular Joint Crepitus
Description: Presence of multiple, distinct joint sounds (crepitus).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | PRGF Arm | Steroid Arm
Number analyzed (Participants) | 4 | 1
Participants | 3 | 0

6. Other Pre Specified Outcome: Temporomandibular Joint Crepitus
Description: Presence of multiple, distinct joint sounds (crepitus).
Time Frame: Six Months
Measure: Count of Participants; unit: Participants
Arm/Group | PRGF Arm | Steroid Arm
Number analyzed (Participants) | 4 | 1
Participants
  TMJ Crepitus Present | 3 | 0
  No TMJ Sound | 1 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | PRGF Arm | Steroid Arm
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1
Other Adverse Events (participants affected / at risk) | 0/4 | 0/1

LIMITATIONS AND CAVEATS:
Due to the limited number of participants in this clinical trial, the study was terminated, and a statistical analysis was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-01-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04731233/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT04731233/SAP_001.pdf